CLINICAL TRIAL: NCT01039727
Title: Prerecorded Autosuggestion in Long-standing Pain Intervention
Acronym: PALPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Free University Medical Center (Other)
Responsible Party: Dr. Jean-Luc Mommaerts, M.D., M.Sc., Free University Brussels
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.U.N. B14320096694
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: Pain [C10.597.617]
MeSH Terms: conditions — Pain | interventions — Compact Disks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- care as usual (No Intervention): care as usual
- autosuggestive support (Experimental): care as usual + 5 specific CDs (3 'General pain relief' + 2 'Short relaxations')
  Interventions: Other: care as usual + 5 specific CDs
- autosuggestive support ++ (Experimental): care as usual + email assistance (password protected) + AurelisOnLine (AoL) + 5 CDs at the start (same as in arm 2) + more CDs as needed after 1 month
  Interventions: Other: care as usual + email assistance + AurelisOnLine (AoL) + CDs

INTERVENTIONS:
Other: care as usual + 5 specific CDs — care as usual + 5 specific CDs (3 'General pain relief' + 2 'Short relaxations')
  Arms: autosuggestive support
Other: care as usual + email assistance + AurelisOnLine (AoL) + CDs — care as usual + email assistance (password protected) + AurelisOnLine (AoL) + 5 CDs at the start (same as in arm 2) + more CDs as needed after 1 month
  Arms: autosuggestive support ++

SUMMARY:
The first objective of this thesis is to investigate the hypothesis that prerecorded autosuggestion (PA) can be a theoretically valuable (efficacy) and practical (efficiency) tool in the care of many patients with chronic pain. With a prevalence in chronic pain conditions of +/- 20% of adults, chronic pain is a huge problem for individuals as well as for society, absorbing an enormous amount of resources. Even with all available treatments, many people still suffer from chronic pain, in particular when this pain has a psychosomatic ('functional') origin. In the PALPI study (Prerecorded Autosuggestion in Long-standing Pain Intervention), accompanying this thesis, efforts are made to mainly involve chronic pain of clearly psychosomatic origin.

DETAILED DESCRIPTION:
A number of GPs will be contacted. A working definition of 'chronic pain patient' is put forward. Only patients with chronic pain for which present research suspects a substantial degree of psychosomatic causality are withheld. A randomization of these into three groups is performed by the appropriate department of the VUB. The three groups are: a control group (receiving 'care as usual'), a group receiving additionally to care as usual, 5 autosuggestion CDs (containing +/- 25 different sessions of autosuggestion) and a group receiving additionally to care as usual, email assistance (through a specific internet module), including downloadable CDs as appropriate and access to 'AurelisOnLine' (an internet application with > 900 different sessions of autosuggestion). Three of the CDs contain pre-recorded sessions of relaxation + autosuggestion aimed at diminishing pain. Other CDs are about relaxation, general wellness, etc. Each arm of investigation contains 30 subjects. Assessments are made at 3 points in time: at the start, at 1 month from the start and at 3 months from the start. The following will be measured: quality of life (through a Dutch version of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI)), levels of pain intensity and quality (through a Dutch version of the McGill Pain Questionnaire (SF-MPQ)) and use of painkillers. In addition to this, the acceptance/satisfaction of physicians and patients of this kind of treatment will also be the subject of this investigation.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged > 18 years.
* The subject is a 'chronic pain patient': at least 3 months of almost daily pain.
* The subject has one of the following syndromes and has been sufficiently investigated upon it in order to exclude a physical medical cause:

  * chronic low back pain
  * chronic thoracic pain
  * chronic neck pain
  * fibromyalgia
  * temporomandibular pain dysfunction (TMPD)
  * complex regional pain syndrome (CRPS) = RSD
  * chronic tension-type headache
  * chronic pelvic pain
  * painful bladder syndrome
  * irritable bowel syndrome
  * vulvodynia
* The subject has a fast internet connection with possibility to download and burn CDs and/or copy mp3s on an mp3-player (or knows someone who is willing to take care of this)
* The subject has a CD and/or mp3 player at disposal or will buy one.

As an additional 'inclusion criterion', we explicitly ask the referring physician to include preferably patients whom he would otherwise also advise PALPI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire - Dutch language Version (MPQ-DLV) | 1 month

SECONDARY OUTCOMES:
Multidimensional Pain Inventory - Dutch language Version (MPI-DLV) | 1 month
Multidimensional Pain Inventory - Dutch language Version (MPI-DLV) | 3 months
McGill Pain Questionnaire - Dutch language Version (MPQ-DLV) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Devroey, Study Chair — Université Libre de Bruxelles
Locations (1):
- Free University Brussels, Brussels, Belgium